CLINICAL TRIAL: NCT07106853
Title: Prenatal Cell-free DNA Screening in Pregnancies With Diverse Genetic Risk Profiles Utilizing Targeted and Whole-exome Sequencing
Status: Not yet recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: University of Pennsylvania (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20250133-R
Record Dates: First submitted 2025-06-11; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, chorionic villus, amniotic cells, cord blood, products of conception (POC), placenta tissues or other tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter study aims to recruit a minimum of 1,600 pregnant women, encompassing individuals with varying levels of genetic risk. The study particularly focuses on cases with increased fetal nuchal translucency (NT ≥3.5 mm), additional ultrasound markers, and/or fetal structural anomalies. Peripheral blood samples of eligible participants will be collected for two state-of-the-art cfDNA tests based on coordinative allele-aware target enrichment sequencing (COATE-seq): (1) a targeted panel to screen for frequent chromosomal aneuploidies, microdeletions/duplications, and dominant single-gene conditions, and (2) comprehensive whole-exome cfDNA sequencing for aneuploidies, microdeletions/duplications, monogenic variants (both dominant and recessive variants), uniparental disomy, and hydatidiform moles. The results of both cfDNA tests will be compared with those from invasive or postnatal diagnostic testing. Pregnancy outcome will be followed up to six weeks postpartum. The primary goal is to determine the clinical validity of targeted and whole exome cfDNA analyses, assessed through sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) relative to diagnostic standards. Secondary goal is to assess efficacy across diverse genetic risk populations by analyzing detection rates of pathogenic variants associated with fetal indications. The clinical utility of cfDNA screening will also be evaluated by its impact on clinical management decisions, including follow-up diagnostic procedures or prenatal/perinatal interventions.

DETAILED DESCRIPTION:
This prospective, multicenter clinical study is designed to evaluate the clinical validity and utility of a novel non-invasive prenatal screening platform, COATE-seq (Coordinative Allele-Aware Target Enrichment Sequencing). The study assesses the performance of cfDNA-based testing that integrates both targeted panel and whole-exome sequencing (WES) approaches to detect a broad range of fetal genetic abnormalities-including aneuploidies, microdeletions, monogenic pathogenic variants, uniparental disomy (UPD), and hydatidiform moles from a single maternal blood sample. The overarching aim is to establish the diagnostic accuracy, clinical effectiveness, and real-world impact of this comprehensive assay in routine prenatal care settings.

The primary objective is to evaluate test performance through standard metrics including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV), benchmarked against confirmatory diagnostic results. The secondary objectives focus on comparing detection rates across genetic risk subgroups (e.g., structural anomalies on ultrasound), quantifying the incremental yield of WES over targeted panels, and assessing clinical impact on management decisions. These endpoints are particularly relevant in an era of expanding therapeutic options for genetic conditions where early, non-invasive detection may significantly influence prenatal or perinatal interventions.

Participants will be pregnant women between 9+0 and 25+6 weeks of gestation with singleton pregnancies who meet the following inclusion criteria:

Age 18 years or older;

Willingness to provide informed consent and participate in all study procedures;

Presence of fetal findings on ultrasound meeting one of the following:

Increased nuchal translucency (NT ≥3.5 mm), with or without additional markers;

Structural anomalies detected on prenatal imaging;

Agreement to undergo at least one molecular diagnostic test (prenatal or postnatal), and possible follow-up testing in family members.

Exclusion criteria include:

Gestational age outside of 9+0 to 25+6 weeks;

Age under 18 years;

Presence of a known familial pathogenic variant fully explaining the fetal ultrasound findings;

Maternal conditions that may confound cfDNA analysis, such as active malignancy, recent allogeneic blood transfusion, organ transplantation, or cell-based therapy within the past year.

The initial visit includes informed consent, demographic and clinical history collection, fetal ultrasound evaluation, and sample collection for cfDNA analysis and diagnostic testing (if available). The cfDNA assay incorporates targeted and exome-based sequencing of fetal DNA fragments isolated from maternal plasma. The second visit is an interim follow-up for review of diagnostic results and patient counseling. The final visit involves pregnancy outcome documentation via chart review or direct follow-up, capturing live birth, miscarriage, stillbirth, or elective termination, and any available postnatal phenotype confirmation.

The COATE-seq assay uses hybrid-capture-based NGS to detect chromosomal aneuploidies (e.g., T21, T18, T13), pathogenic microdeletions (e.g., 22q11.2 deletion syndrome), and a curated panel of 56 monogenic conditions selected through the SEPH framework prioritizing severe, early-onset, prevalent, and analytically detectable disorders. The complementary WES component targets ~19,000 genes to broaden detection beyond predefined panels and support exploratory analysis of novel or rare variants. Variant interpretation adheres to ACMG guidelines, and only pathogenic or likely pathogenic variants associated with serious outcomes are reported.

All cfDNA results are compared against one or more reference diagnostic methods, including karyotyping, chromosomal microarray (CMA), targeted gene panels, WES, and whole-genome sequencing. In selected cases, UPD is confirmed via methylation-specific testing or STR profiling. Performance metrics will be calculated on subjects with completed cfDNA and diagnostic data, and efficacy analyses will examine detection rates by condition type and risk strata. Quality assurance measures are built into all stages of the protocol, from sample collection and transport to bioinformatic analysis and reporting.

This study complies with Good Clinical Practice (GCP) and all relevant ethical regulations. Institutional Review Board (IRB) approval is required at each participating site, and informed consent is obtained prior to any study procedures. Confidentiality of subject data is strictly maintained, and adverse events including complications from invasive diagnostic procedures. The study's findings will be disseminated via scientific publications and presentations, contributing to the evidence base for expanded cfDNA screening in prenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant woman (≥18 years old)
* Gestational age between 9+0 and 25+6 weeks
* Singleton pregnancy
* Pregnancy with indications for prenatal diagnosis due to:

  * Increased nuchal translucency (NT) ≥3.5 mm: capped at 25% of total subjects
  * Increased NT ≥3.5 mm AND presence of any other "soft marker" or structural anomaly: capped at 25% of total subjects
  * Presence of structural anomaly: at least 50% of total subjects
* Agree to participate in the clinical study for being followed-up and accept at least one molecular diagnosis (diagnostic procedures performed on prenatal invasive specimens, product of conception, umbilical cord blood, or other specimens) and possible family member testing

Exclusion Criteria:

* Age under 18 years
* Gestational age is less than 9+0 weeks or greater than 25+6 weeks
* One parent or other family member has a known pathogenic variant linked to the fetal ultrasound finding(s)
* Conditions affecting the accuracy of cfDNA assay (e.g., maternal malignancy during pregnancy, maternal allogeneic blood transfusion, organ transplantation, or cell therapy within the past year)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: * Adult pregnant woman (≥18 years old)
  * Gestational age between 9+0 and 25+6 weeks
  * Singleton pregnancy
  * Pregnancy with indications for prenatal diagnosis due to:
    * Increased nuchal translucency (NT) ≥3.5 mm: capped at 25% of total subjects
    * Increased NT ≥3.5 mm AND presence of any other "soft marker" or structural anomaly: capped at 25% of total subjects
    * Presence of structural anomaly: at least 50% of total subjects
  * Agree to participate in the clinical study for being followed-up and accept at least one molecular diagnosis (diagnostic procedures performed on prenatal invasive specimens, product of conception, umbilical cord blood, or other specimens) and possible family member testing
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Determine the clinical validity of targeted and whole exome cfDNA analyses, assessed through sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) relative to diagnostic standards. | 18 months

SECONDARY OUTCOMES:
Assess efficacy across diverse genetic risk populations by analyzing detection rates of pathogenic variants associated with fetal indications. | 8 months

IPD SHARING:
Plan to Share IPD: Yes
IPD will be part of the data published for the study results.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD will be available together with the publication of the study results.